CLINICAL TRIAL: NCT06011005
Title: Efficacy of Ethyl Chloride Topical Anesthesia Application on the Pain Perception During Intra-oral Injections in Children in Comparison to Benzocaine Gel- a Single-blinded Randomized Controlled Trial.
Brief Title: Efficacy of Ethyl Chloride Topical Anesthesia Application on the Pain Perception During Intra-oral Injections in Children in Comparison to Benzocaine Gel.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Nagah ABdelrahman, Principal Investigator, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MBRU IRB-2022-174
Record Dates: First submitted 2023-07-05; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Dental Caries in Children; Anesthesia, Local; Injection Site Discomfort

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group A) Ethyl Chloride (EC) (Experimental): Topical application for 30 sec.
  Interventions: Other: Ethyl Chloride spray (group A)
- (Group B) Benzocaine gel 20% (BC) (Active Comparator): BC 20% Topical gel application for 30 sec and left for 1 minute.
  Interventions: Other: Benzocaine gel 20% (group B)

INTERVENTIONS:
Other: Ethyl Chloride spray (group A) — Cold test spray
  Arms: (Group A) Ethyl Chloride (EC)
Other: Benzocaine gel 20% (group B) — Topical analgesia
  Arms: (Group B) Benzocaine gel 20% (BC)

SUMMARY:
The goal of this single-blinded randomized controlled trial is to compare pain perception during buccal infiltration using indirect EC spray and topical anesthesia and BC 20% topical gel, among seven to 10-year-old school children who attended Pediatric Dentistry Department at Dubai Dental Hospital (DDH), Mohammed Bin Rashid University (MBRU) in Dubai, the United Arab Emirates (UAE).

The main question[s] it aims to answer are:

• How effective is the indirect application of EC topical spray anesthesia on pain perception during intraoral buccal injection in children in comparsion to BC 20%?

Researchers will compare efficacy of 20% Benzocaine (BC) gel and indirect application of Ethyl Chloride (EC) spray to see if reducing pain perception during local anesthesia infiltration.

DETAILED DESCRIPTION:
Pre-local analgesia topical Benzocaine gel or Ethyl Chloride technique will be selected randomly and applied per the protocol. A single calibrated operator (A.A) using randomly selected sealed envelopes that have been previously divided equally according to sample size arms. The selected envelope is then opened by the operator, who applies either the EC or BC topical anesthesia technique based on the chosen envelop. Followed by maxillary local analgesia buccal infiltration for a single tooth by a calibrated operator (A.A). The child is then observed and assessed by the blinded primary investigator (N.A) (to the topical anesthesia technique) for pain perception during local anesthesia infiltration based on the Sound, Eye, Motor index used in this study. The child is then asked to rate the Visual Analog Scale and Facial Pain Scale. Heart rate of the patient will be recorded as per below protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (ASA I) aged between 7 - 10 years old.
* Needing any maxillary buccal infiltration (anterior, middle, posterior)
* Had no prior history of local anesthesia.
* Frankl behavior III or IV
* Not taking any painkillers, or other drugs that would influence with their pain perception.

Exclusion Criteria:

* History of a medically compromised condition and intellectual disability. § Any allergy to local anesthesia.
* Active pathology at the site of injection.
* Prior history of intra-oral injection.
* Frankl behavior I or II.
* Children/parents not willing to participate in the study. § Needle phobia.
* Patients require treatment under conscious sedation.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-10-24 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate | 5-10 minutes
  Each participant's heart rate will be recorded immediately before and after the injection using an FDA-approved pulse oximeter.

SECONDARY OUTCOMES:
Sound, Eye, Motor (SEM) Index | 5-10 minutes
  During the insertion of the needle, the operator will evaluate the patient's behavior for pain perception using sound, eye, motor (SEM) scale and visual analog scale (VAS).
Visual Analog Scale (VAS) | 5-10 minutes
  The VAS scale is a 100-mm long horizontal line labeled "no pain: at one end and "worst pain possible" at the other. After each procedure (EC or BC), the participants are asked to evaluate the degree of pain (primary outcome) they experienced using the Facial Pain Scale below.
Face Pain Scale | 5-10 minutes
  These faces show how much something can hurt. This face (point to leftmost face] shows no pain. The faces show more and more pain [point to each from left to the right] up to this one [point to rightmost face] - it shows very much pain. Point to the face that shows how much the child is hurt. Score the chosen face 0, 2, 4, 6, 8, or 10, counting left to right, so ''0' = 'no pain' and ''10' = 'very much pain. Do not use words like "happy' and ''sad'. This scale is intended to measure how children feel inside, not how their face looks. Brief word instructions: Point to each face using the words to describe the pain intensity. Ask the children to choose a face that best describes their pain and record the appropriate number.

CONTACTS AND LOCATIONS:
Overall Officials: Nagah Abdelrahman, Principal Investigator — Mohammed Bin Rashid University of Medicine and Health Sciences
Locations (1):
- Mohammed Bin Rashid University Of Medicine and Health Sciences, Multiple Locations, United Arab Emirates

REFERENCES:
- [Result] Dasarraju RK, Svsg N. Comparative efficacy of three topical anesthetics on 7-11-year-old children: a randomized clinical study. J Dent Anesth Pain Med. 2020 Feb;20(1):29-37. doi: 10.17245/jdapm.2020.20.1.29. Epub 2020 Feb 28. PMID 32158957
- [Result] Lakshmanan L, Ravindran V. Efficacy of Cryotherapy Application on the Pain Perception during Intraoral Injection: A Randomized Controlled Trial. Int J Clin Pediatr Dent. 2021 Sep-Oct;14(5):616-620. doi: 10.5005/jp-journals-10005-2032. PMID 34934271
- [Result] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Result] Kreider KA, Stratmann RG, Milano M, Agostini FG, Munsell M. Reducing children's injection pain: lidocaine patches versus topical benzocaine gel. Pediatr Dent. 2001 Jan-Feb;23(1):19-23. PMID 11242725
- [Result] Gill CJ, Orr DL 2nd. A double-blind crossover comparison of topical anesthetics. J Am Dent Assoc. 1979 Feb;98(2):213-4. doi: 10.14219/jada.archive.1979.0476. PMID 370178
- [Result] Lathwal G, Pandit IK, Gugnani N, Gupta M. Efficacy of Different Precooling Agents and Topical Anesthetics on the Pain Perception during Intraoral Injection: A Comparative Clinical Study. Int J Clin Pediatr Dent. 2015 May-Aug;8(2):119-22. doi: 10.5005/jp-journals-10005-1296. Epub 2015 Aug 11. PMID 26379379
- [Result] Hindocha N, Manhem F, Backryd E, Bagesund M. Ice versus lidocaine 5% gel for topical anaesthesia of oral mucosa - a randomized cross-over study. BMC Anesthesiol. 2019 Dec 16;19(1):227. doi: 10.1186/s12871-019-0902-8. PMID 31842771
- [Result] Hersh EV, Houpt MI, Cooper SA, Feldman RS, Wolff MS, Levin LM. Analgesic efficacy and safety of an intraoral lidocaine patch. J Am Dent Assoc. 1996 Nov;127(11):1626-34; quiz 1665-6. doi: 10.14219/jada.archive.1996.0098. PMID 8952239
- [Result] Amado A, Sood A, Taylor JS. Contact allergy to lidocaine: a report of sixteen cases. Dermatitis. 2007 Dec;18(4):215-20. doi: 10.2310/6620.2007.06059. PMID 18021602
- [Result] Silver K, Silver J. The place of James Arnott (1797-1883) in the development of local anaesthesia in dentistry. Br Dent J. 2016 Mar 11;220(5):249-52. doi: 10.1038/sj.bdj.2016.179. PMID 26964600
- [Result] Davoudi A, Rismanchian M, Akhavan A, Nosouhian S, Bajoghli F, Haghighat A, Arbabzadeh F, Samimi P, Fiez A, Shadmehr E, Tabari K, Jahadi S. A brief review on the efficacy of different possible and nonpharmacological techniques in eliminating discomfort of local anesthesia injection during dental procedures. Anesth Essays Res. 2016 Jan-Apr;10(1):13-6. doi: 10.4103/0259-1162.167846. PMID 26957683
- [Result] Ernst E, Fialka V. Ice freezes pain? A review of the clinical effectiveness of analgesic cold therapy. J Pain Symptom Manage. 1994 Jan;9(1):56-9. doi: 10.1016/0885-3924(94)90150-3. PMID 8169463
- [Result] Malanga GA, Yan N, Stark J. Mechanisms and efficacy of heat and cold therapies for musculoskeletal injury. Postgrad Med. 2015 Jan;127(1):57-65. doi: 10.1080/00325481.2015.992719. Epub 2014 Dec 15. PMID 25526231
- [Result] Kosaraju A, Vandewalle KS. A comparison of a refrigerant and a topical anesthetic gel as preinjection anesthetics: a clinical evaluation. J Am Dent Assoc. 2009 Jan;140(1):68-72; quiz 112-3. doi: 10.14219/jada.archive.2009.0020. PMID 19119169
- [Result] DiMarco AC, Wetmore AO. Clinical Comparison: Fast-Acting and Traditional Topical Dental Anesthetic. Anesth Prog. 2016 Summer;63(2):55-61. doi: 10.2344/0003-3006-63.2.55. PMID 27269661
- [Result] Ballesteros-Pena S, Fernandez-Aedo I, Vallejo-De la Hoz G; en representacion del Grupo de Trabajo DIASURE. [Ethyl chloride aerosol spray for local anesthesia before arterial puncture: randomized placebo-controlled trial]. Emergencias. 2017 Jun;29(3):161-166. Spanish. PMID 28825235
- [Result] French JO, Hooker ML, Vause RB, Robinson AL. Dental Anaesthesia in Children: A Comparison of Vinyl Ether and Ethyl Chloride. Br Med J. 1940 Mar 16;1(4132):432-5. doi: 10.1136/bmj.1.4132.432. No abstract available. PMID 20783002
- [Result] Hori A, Poureslami HR, Parirokh M, Mirzazadeh A, Abbott P. The ability of pulp sensibility tests to evaluate the pulp status in primary teeth. Int J Paediatr Dent. 2011 Nov;21(6):441-5. doi: 10.1111/j.1365-263X.2011.01147.x. Epub 2011 Jun 27. PMID 21702853
- [Result] Asfour MA, Millar BJ, Smith PB. An assessment of the reliability of pulp testing deciduous teeth. Int J Paediatr Dent. 1996 Sep;6(3):163-6. doi: 10.1111/j.1365-263x.1996.tb00235.x. PMID 9115971
- [Result] Russell SC, Doyle E. A risk-benefit assessment of topical percutaneous local anaesthetics in children. Drug Saf. 1997 Apr;16(4):279-87. doi: 10.2165/00002018-199716040-00005. PMID 9113495
- Available data/document: Study Protocol: MBRU IRB-2022-174 — http://www.mbru.ac.ae

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT06011005/Prot_SAP_ICF_000.pdf